CLINICAL TRIAL: NCT01760577
Title: Comparing Effects of Intraarticular Botulinum Toxin A Versus Hyaluronate Plus Rehabilitation Exercise in Patients With Unilateral Ankle Osteoarthritis
Brief Title: Effects of Intraarticular Botulinum Toxin A in Ankle Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Shu-Fen Sun, MD, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VGHKS100-061
Record Dates: First submitted 2012-12-30; First posted 2013-01-04 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Ankle Osteoarthritis
Keywords: osteoarthritis, botulinum toxin, hyaluronate
MeSH Terms: conditions — Osteoarthritis | interventions — Botulinum Toxins, Type A; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The Botulinum Toxin A group (Experimental): The Botulinum Toxin A group received intraarticular injections of 100 units of Botulinum Toxin A (Allergan, Inc, Irvine CA) reconstituted in 2 cc normal saline.
  Interventions: Drug: Botulinum Toxin A (Allergan, Inc, Irvine CA)
- The hyaluronate group (Hyalgan, Italy) (Active Comparator): The hyaluronate group received intraarticular injections of 2 ml sodium hyaluronate (Hyalgan, molecular weight 500-730kDa, Fidia Pharmaceutical Corporation, Abano Terme, Italy) and subsequent 6 sessions of rehabilitation exercise for 50 miniutes/day, 3 days per week for 2 weeks and home exercise for 2 weeks .
  Interventions: Drug: Hyalgan (Hyalgan, Fidia , Italy)

INTERVENTIONS:
Drug: Botulinum Toxin A (Allergan, Inc, Irvine CA) — patients received intraarticular injections by the same experienced physician using aseptic procedures.
  Other Names: 100 units of Botulinum Toxin A in 2 cc NS
  Arms: The Botulinum Toxin A group
Drug: Hyalgan (Hyalgan, Fidia , Italy) — The rehabilitation program consists of 6 sessions of rehabilitation exercise for 50 miniutes/day, 3 days per week for 2 weeks and home exercise program for another 2 weeks.
  Other Names: 2 ml Hyalgan, molecular weight 500-730kDa, Fidia , Italy
  Arms: The hyaluronate group (Hyalgan, Italy)

SUMMARY:
The purpose of this study is to compare the effects of intraarticular Botulinum Toxin A versus intraarticular hyaluronate plus rehabilitation exercise in patients with ankle osteoarthritis.

DETAILED DESCRIPTION:
Recent pilot studies report that intraarticular injection of Botulinum Toxin A into painful joints of patients with various types of arthritis leads to significant and durable improvement in pain and function and is safe to use. To date, there is no published literature that evaluate the effects of intraarticular Botulinum Toxin A in the treatment of ankle OA. Sun el al reported that 3 or 5 weekly injection of hyaluronate may improve pain and physical function in patients with ankle OA and the treatment effects may last for 6 months. The effect of one injection of hyaluronate plus exercise had never been studied. The purpose of this study is to compare the effects of intraarticular Botulinum Toxin A versus intraarticular hyaluronate plus rehabilitation exercise for patients with ankle OA.

ELIGIBILITY:
Inclusion Criteria:

* an age of 20-85 years with diagnosis of ankle osteoarthritis
* unilateral ankle pain that had lasted for at least 6 months, with no significant benefit from conservative treatment or with an inability to tolerate the side effects of medications
* ankle radiographs taken within 6 months equivalent to grade 2 on the Kellgren-Lawrence grading system
* a current total Ankle Osteoarthritis Scale (AOS) score of >3 and < 9 (possible range, 0-10)
* a normal activity level-i.e., not bedridden or confined to a wheelchair, and are able to walk 30 meters without the aid of a walker, crutches or cane
* no changes in shoes or orthotic devices during the study period.

Exclusion Criteria:

* pregnancy or lactation in women
* lower leg trauma other than ankle trauma
* previous surgery involving the spine, hip or knee
* the presence of an active joint infections of foot or ankle
* previous surgery or arthroscopy on the ankle within 12 months
* history of chicken or egg allergy
* intraarticular steroid or hyaluronate injection in the treated ankle within the previous 6 months
* treatment with anticoagulants or immunosuppressives
* a history of rheumatoid arthritis, gout, or any other inflammatory arthropathy
* the presence of other comorbidity (such as neoplasms, diabetes mellitus, paresis or recent trauma) or poor health status that would interfere with the clinical assessments during the study.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-05; Primary Completion 2012-05 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Ankle Osteoarthritis Scale (AOS) score | at 6 months after the injection
  The AOS is a patient-rated, validated outcome measure that includes nine items on a pain subscale and nine items on a disability subscale.Using the AOS, a score of 0 represent no pain or disability and 10 represent worst pain or disability imaginable

SECONDARY OUTCOMES:
AOFAS ankle/hindfoot score | pre-injection and at 2 weeks, 1 month, 3 months, and 6 months post injection.
  AOFAS ankle/hindfoot score is a 100-point scale that devotes 40 points to pain, 50 points to function and 10 points to alignment.
Visual analog scale (VAS) | pre-injection and at 2 weeks, 1 month, 3 months, and 6 months post injection
  The patient rate the intensity of average ankle movement pain in the previous week using a 10-cm horizontal Visual analog scale (VAS)
Single-leg stance test (SLS) | pre-injection and at 2 weeks, 1 month, 3 months, and 6 months post injection
  Single-leg stance test (SLS) is done by raising one foot up without touching it to the supported lower extremity with ankle OA and maintain balance for as long as possible
Timed " Up-and-Go" test (TUG) | pre-injection and at 2 weeks, 1 month, 3 months, and 6 months post injection
  A Timed " Up-and-Go" test (TUG) measures functional mobility and the dynamic balance of an individual.
global Patients satisfaction | at 2 weeks, 1 month, 3 months, and 6 months post injection.
  This rating is based on a 7-point categorical scale ranging from completely satisfied, satisfied, somewhat satisfied, no change, somewhat unsatisfied, unsatisfied to completely unsatisfied.
adverse effects | at 2 weeks, 1 month, 3 months, and 6 months post injection.
  patients recorded any systemic and local adverse effects (defined as any unwanted effect whether it was thought to be related to the study or not) on a diary card.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Fen Sun, MD, Principal Investigator — Kaohsiung Veterans General Hospital, Taiwan
Locations (1):
- Kaohsiung Veterans General Hospital, No 386, Ta-Chung 1st Road, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Sun SF, Chou YJ, Hsu CW, Hwang CW, Hsu PT, Wang JL, Hsu YW, Chou MC. Efficacy of intra-articular hyaluronic acid in patients with osteoarthritis of the ankle: a prospective study. Osteoarthritis Cartilage. 2006 Sep;14(9):867-74. doi: 10.1016/j.joca.2006.03.003. Epub 2006 Apr 24. PMID 16635582
- [Background] Sun SF, Hsu CW, Sun HP, Chou YJ, Li HJ, Wang JL. The effect of three weekly intra-articular injections of hyaluronate on pain, function, and balance in patients with unilateral ankle arthritis. J Bone Joint Surg Am. 2011 Sep 21;93(18):1720-6. doi: 10.2106/JBJS.J.00315. PMID 21938376
- [Background] Mahowald ML, Singh JA, Dykstra D. Long term effects of intra-articular botulinum toxin A for refractory joint pain. Neurotox Res. 2006 Apr;9(2-3):179-88. doi: 10.1007/BF03033937. PMID 16785116
- [Background] Singh JA, Mahowald ML, Kushnaryov A, Goelz E, Dykstra D. Repeat injections of intra-articular botulinum toxin a for the treatment of chronic arthritis joint pain. J Clin Rheumatol. 2009 Feb;15(1):35-8. doi: 10.1097/RHU.0b013e3181953b14. No abstract available. PMID 19131763
- [Background] Singh JA, Mahowald ML, Noorbaloochi S. Intra-articular botulinum toxin A for refractory shoulder pain: a randomized, double-blinded, placebo-controlled trial. Transl Res. 2009 May;153(5):205-16. doi: 10.1016/j.trsl.2009.02.004. Epub 2009 Mar 13. PMID 19375681
- [Background] Mahowald ML, Krug HE, Singh JA, Dykstra D. Intra-articular Botulinum Toxin Type A: a new approach to treat arthritis joint pain. Toxicon. 2009 Oct;54(5):658-67. doi: 10.1016/j.toxicon.2009.03.028. Epub 2009 Apr 5. PMID 19351542
- [Background] Aoki KR. Evidence for antinociceptive activity of botulinum toxin type A in pain management. Headache. 2003 Jul-Aug;43 Suppl 1:S9-15. doi: 10.1046/j.1526-4610.43.7s.3.x. PMID 12887389
- [Background] Sun SF, Chou YJ, Hsu CW, Chen WL. Hyaluronic acid as a treatment for ankle osteoarthritis. Curr Rev Musculoskelet Med. 2009 Jun;2(2):78-82. doi: 10.1007/s12178-009-9048-5. Epub 2009 Mar 13. PMID 19468874
- [Background] Konttinen YT, Kemppinen P, Segerberg M, Hukkanen M, Rees R, Santavirta S, Sorsa T, Pertovaara A, Polak JM. Peripheral and spinal neural mechanisms in arthritis, with particular reference to treatment of inflammation and pain. Arthritis Rheum. 1994 Jul;37(7):965-82. doi: 10.1002/art.1780370701. No abstract available. PMID 8024624
- [Derived] Sun SF, Hsu CW, Lin HS, Chou YJ, Chen JY, Wang JL. Efficacy of intraarticular botulinum toxin A and intraarticular hyaluronate plus rehabilitation exercise in patients with unilateral ankle osteoarthritis: a randomized controlled trial. J Foot Ankle Res. 2014 Feb 6;7(1):9. doi: 10.1186/1757-1146-7-9. PMID 24502534